CLINICAL TRIAL: NCT04297462
Title: Efficacy of Different Regimens in Influenza Postexposure Chemoprophylaxis With Oral Neuraminidase Inhibitor in Children
Brief Title: Different Regimens in Influenza Postexposure Chemoprophylaxis in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, August Wrotek, Principal Investigator, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 77/PB/2016
Record Dates: First submitted 2020-02-18; First posted 2020-03-05 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Influenza; Exposure; Prevention
Keywords: influenza; chemoprevention; oseltamivir; child; infant
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Intervention Model Description: Patients randomly allocated into 3 or 7-days postexposure chemoprophylaxis group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-days postexposure chemoprophylaxis (Experimental): Oseltamivir given orally, 3mg per each body kg, once a day during three consecutive days after the contact with influenza
  Interventions: Drug: Oseltamivir 3 days
- 7-days postexposure chemoprophylaxis (Active Comparator): Oseltamivir given orally, 3mg per each body kg, once a day during seven consecutive days after the contact with influenza
  Interventions: Drug: Oseltamivir 7 days

INTERVENTIONS:
Drug: Oseltamivir 3 days — Non-inferiority study of 3 versus 7-days duration of PEP
  Other Names: 3-days postexposure chemoprophylaxis with oseltamivir
  Arms: 3-days postexposure chemoprophylaxis
Drug: Oseltamivir 7 days — Active comparator
  Other Names: 7-days postexposure chemoprophylaxis with oseltamivir
  Arms: 7-days postexposure chemoprophylaxis

SUMMARY:
Although the vaccination is the preferred method of influenza prevention, there are some occasions on which a postexposure prophylaxis (PEP) is required. Two neuraminidase inhibitors (NAIs) may be used in chemoprophylaxis in children: oral oseltamivir, and inhaled zanamivir. Both, oseltamivir and zanamivir, are effective in treatment and in prophylaxis of influenza, and the efficacy is calculated to reach 70-90%. Oseltamivir is used more frequently, since zanamivir is licensed in older children (5 years of age and above), and children under the age of 5 years are at higher risk of influenza complications. Oseltamivir use correlated in children with higher risk of vomiting, with no increased risk of other adverse events, including those observed in adult patients (nausea, renal events, and psychiatric effects). The PEP may be indicated by individual patient's characteristics (e.g. patients in high-risk group) or epidemiological reasons, i.e. prevention of institutional outbreaks.The one research that analyzed efficacy of 3-days PEP versus 7 or 10-days and showed overall efficacy of shorter oseltamivir prophylaxis to be high and comparable to that of longer regimens. The study included several pediatric patients and made the investigators perform such an analysis in pediatric population. In this randomized controlled trial, the investigators aimed to compare efficacy, safety, and costs of 3 versus 7-days prophylaxis with oral oseltamivir in children hospitalized. The hypothesis is that 3-days duration of PEP is not less effective than 7-days PEP, and patients might gain from lower number of adverse reactions related to drug administration.

DETAILED DESCRIPTION:
Only applies to patients hospitalized due to other than influenza reasons. If a proven contact with influenza has taken place (influenza diagnosed by signs/symptoms and positive rapid influenza diagnostic test and/or PCR), a patient may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized at the Pediatric Ward
* age: 0-18 years old
* confirmed contact with a person diagnosed with influenza
* patient's, patient's parent/tutor's informed consent

Exclusion Criteria:

* lack of an informed consent
* more than 48 hours after the first contact with influenza
* severe adverse reaction to the drug- discontinuation of the prophylaxis
* important to a parent/tutor drug intolerance (e.g. lack of tolerance of a drug's taste)
* new contact with influenza after chemoprophylaxis has finished

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Postexposure chemoprophylaxis efficacy | up to 7 days after PEP has finished
  Percent of patients who did not have influenza in each study arm.
Oseltamivir safety | up to 7 days after PEP has finished
  Presence of the following adverse reactions to drug (in percents): nausea, vomiting, skin hypersensitivity (including rash), sleep disorders, consciousness disorders, convulsions, fever related to drug administration, symptomatic arrhythmias, behavioral changes
Postexposure chemoprophylaxis costs | up to 7 days after PEP has finished
  Cost of drugs used in each arm, costs of treatment of adverse reactions

SECONDARY OUTCOMES:
Need for hospitalization in case of influenza after failed chemoprophylaxis | Up to 28 days
  A need for hospitalization if influenza is present within 7 days after PEP completion
Duration of influenza signs and symptoms after failed chemoprophylaxis | Up to 28 days
  Length of period when signs and symptoms are present
Presence of complications in case of influenza after failed chemoprophylaxis | Up to 28 days
  Presence of influenza complications: pneumonia, bronchitis, otitis media, need for antibiotic treatment, neurological sequelae, ICU transfer, death
Fever in case of influenza after failed chemoprophylaxis | Up to 28 days
  Highest fever and duration of fever

CONTACTS AND LOCATIONS:
Overall Officials: August E. Wrotek, MD PhD, Principal Investigator — The Centre of Postgraduate Medical Education
Locations (1):
- The Centre of Postgraduate Medical Education, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Background] Ishiguro N, Oyamada R, Nasuhara Y, Yamada T, Miyamoto T, Imai S, Akizawa K, Fukumoto T, Iwasaki S, Iijima H, Ono K. Three-day regimen of oseltamivir for postexposure prophylaxis of influenza in wards. J Hosp Infect. 2016 Oct;94(2):150-3. doi: 10.1016/j.jhin.2016.05.012. Epub 2016 May 25. PMID 27346624
- [Derived] Wrotek A, Jackowska T. A noninferiority randomized open-label pilot study of 3- versus 7-day influenza postexposure prophylaxis with oseltamivir in hospitalized children. Sci Rep. 2024 Jun 20;14(1):14192. doi: 10.1038/s41598-024-65244-5. PMID 38902383
- See also: Three-day regimen of oseltamivir for postexposure prophylaxis of influenza in wards. — https://www.ncbi.nlm.nih.gov/pubmed/?term=ishiguro+postexposure